CLINICAL TRIAL: NCT04364620
Title: A Phase II Study of AB-16B5 Combined With Docetaxel in Previously Treated Subjects With Metastatic Non-Small Cell Lung Cancer (EGIA-002)
Brief Title: AB-16B5 Combined With Docetaxel in Subjects With Metastatic Non-Small Cell Lung Cancer (EGIA-002)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alethia Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AB-16B5-201
Record Dates: First submitted 2020-04-23; First posted 2020-04-28 (Actual); Results first posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: NSCLC Stage IV
Keywords: Lung cancer; Chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Docetaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm AB-16B5 and Docetaxel (Experimental): AB-16B5 at a dose of 12 mg/kg once weekly on Days 1, 8 and 15 combined with docetaxel at a dose of 75 mg/m2 once every 3 weeks on Day 1.
  Interventions: Drug: AB-16B5; Drug: Docetaxel

INTERVENTIONS:
Drug: AB-16B5 — AB-16B5 is an inhibitor of the epithelial to mesenchymal transition. It is a fully humanized monoclonal antibody of IgG2 isotype against tumor-associated secreted clusterin (TA-sCLU).
Drug: Docetaxel — Docetaxel is an anticancer chemotherapy drug approved in the treatment of non-small cell lung cancer

SUMMARY:
This Phase II study will recruit 40 metastatic non-small cell lung cancer patients who failed treatment with a platinum-containing doublet treatment and an anti-PD1 or PD-L1 immune checkpoint antibody, administered simultaneously or sequentially. All recruited patients will receive AB-16B5 at a dose of 12 mg/kg once weekly combined with docetaxel at a dose of 75 mg/m2 once every 3 weeks.

DETAILED DESCRIPTION:
This is an open-label, single-arm, multi-center Phase II trial of AB-16B5 in combination with docetaxel in previously treated subjects with metastatic non-small cell lung cancer who have experienced disease progression following treatment with a platinum-containing doublet treatment and an anti-PD1 or PD-L1 immune checkpoint antibody, administered simultaneously or sequentially. Approximately 40 subjects will be enrolled in this trial and receive AB-16B5 at a dose of 12 mg/kg once weekly on Days 1, 8 and 15 combined with docetaxel at a dose of 75 mg/m2 once every 3 weeks on Day 1. One cycle of treatment will consist of 21 days (3 weeks). The safety profile of the AB-16B5 and docetaxel combination will be examined during a safety lead-in period with the first 8 subjects completing one cycle of treatment. No dose escalation will be performed but a decision to de-escalate the AB-16B5 dose could be made using the modified toxicity probability interval method.

Subjects will be evaluated every 6 weeks with radiographic imaging to assess response to treatment using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria for determination of the objective response rate (ORR) and progression free survival (PFS). Paired tumor biopsies (pre-treatment and on-treatment) will be collected in all subjects. Study treatment will continue until there is evidence of disease progression, treatment-related adverse events of unacceptable severity, subject request for discontinuation or Investigator determination that further treatment is not in the subject's best interest. Treatment through progression will be allowed if the Investigator considers the subject to be clinically stable. Subjects who must discontinue docetaxel due to toxicity will continue on AB-16B5.

ELIGIBILITY:
Inclusion Criteria:

* Subjects (male or non-pregnant female) must be ≥ 18 years of age on the day of signing the informed consent.
* Subjects with a histologically or cytologically confirmed diagnosis of (Stage III-IV) non-small cell lung cancer (NSCLC) and with at least one measurable lesion defined by RECIST 1.1.
* Subjects must have experienced a disease progression following treatment with an anti-PD1 or PD-L1 immune checkpoint antibody and a platinum-containing doublet treatment, administered simultaneously or sequentially.
* Subjects with a targetable driver mutation in EGFR or ALK gene will be allowed on trial after failing all available targeted therapies and having experienced a disease progression following treatment with an anti-PD1 or PD-L1 immune checkpoint antibody and a platinum-containing doublet treatment, administered simultaneously or sequentially.
* Subjects must have adequate organ and immune function
* Subjects must have a tumor lesion amenable for biopsies with no contraindication for biopsy.
* Subjects must have an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2.
* Subjects must have a life expectancy of at least 3 months.
* Subjects must have recovered from the toxic effects resulting from the most recent cancer treatment to Grade 1 or less. If the subjects underwent major surgery or received radiation therapy, they must have recovered from the complications and/or toxicity.
* Female subjects of childbearing potential must have a negative serum pregnancy test within 72 hours prior to the first dose of study treatment.
* Subjects (both male and female) of reproductive potential must be willing to practice highly effective methods of contraception throughout the study and for up to 90 days after the last dose of study medication. Abstinence is acceptable if this is the subject's usual lifestyle.
* Female subjects are not considered of childbearing potential if they have a history of surgical sterility or evidence of post-menopausal status defined as any of the following:

  * ≥ 45 years of age and has not had menses for more than 2 years.
  * Amenorrhoeic for less than 2 years without hysterectomy and oophorectomy and a follicle stimulating hormone (FSH) value in the postmenopausal range at screening.
  * Post hysterectomy, oophorectomy or tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or by ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure.
* Subjects must understand and be able and willing and likely to fully comply with the study procedures, including scheduled follow-up, and restrictions.
* Subjects must have given written personally signed and dated informed consent to participate in the study in accordance with the International Conference on Harmonization (ICH) Good Clinical Practice (GCP) Guidelines, before completing any study related procedures.

Exclusion Criteria:

* Subjects who have received prior therapy with AB-16B5.
* Subjects who have received prior therapy with docetaxel for the treatment of NSCLC.
* Subjects who are currently participating or has participated in a study of an investigational agent or using an investigational device within 21 days prior to the first dose of study treatment. The 21-day window should be calculated using the last dose of an antineoplastic investigational agent or last use of an investigational device with antineoplastic intent.
* Subjects who have received any anti-cancer treatment within 3 weeks or radiation therapy within 2 weeks prior to receiving the first dose of study treatment or who have not recovered from adverse events to Grade 1 or less. Subjects with alopecia are eligible to participate.
* Subjects who are expected to require any other form of systemic or localized antineoplastic therapy while on the trial. This includes maintenance therapy with another agent or radiation therapy.
* Subjects who are receiving a dose > 10 mg/day of prednisone (or equivalent) within 7 days prior to the first dose of study treatment or any other form of immunosuppressive medication (corticosteroid pre-treatment and/or post-treatment of docetaxel is allowed).
* Subjects who require treatment with a strong CYP3A4 inhibitor (e.g., ketoconazole, itraconazole, clarithromycin, atazanavir, indinavir, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin and voriconazole). Subjects may be included if there is an alternate treatment with a weak CYP3A4 inhibitor and they are willing to change at least 7 days prior to the first dose of study treatment.
* Subjects who have another malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin or in situ cervical cancer.
* Subjects who have known active central nervous system metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate if they have been clinically stable for at least 2 weeks prior to the first dose of study treatment, if they have no evidence of new or enlarging brain metastases and if they are not receiving a dose > 10 mg/day of prednisone (or equivalent) within 7 days prior to the first dose of study treatment.
* Subjects with clinically significant ECG abnormalities.
* Subjects who have received or will receive a live vaccine within 30 days prior to the first dose of study treatment.
* Subjects with a known history of human immunodeficiency (HIV).
* Subjects with an active Hepatitis B or C infection.
* Subjects with an active infection requiring antibiotic therapy.
* Subjects with a known history of alcohol or other substance abuse within the last year.
* Subjects with known hypersensitivity to docetaxel.
* Subjects who have a history or current evidence of any condition, therapy or laboratory abnormalities that may confound the results of the trial, interfere with the subject's participation for the full duration of the trial or if it is not in the best interest of the subject to participate in the trial.
* Subjects with medical, social or psychosocial factors that, in the opinion of the treating Investigator, could impact the safety or compliance with study procedures.
* Subjects who are pregnant or lactating or who are expecting to conceive or father children within the projected duration of the trial through 90 days after the last dose of AB-16B5 or the last dose of docetaxel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Laurin, Study Director — Alethia Biotherapeutics Inc.
Locations (5):
- The University of Texas MD Anderson Cancer Center, Houston, Texas, United States
- Canada (4):
  - Hôpital Maisonneuve-Rosemont, Montreal, Quebec
  - Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec (IUCPQ), Québec, Quebec
  - Centre Intégré de Santé et de Services Sociaux des Laurentides (Hôpital Régional de St-Jérôme), Saint-Jérôme, Quebec

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- AB-16B5 12 mg/kg & Docetaxel 75 mg/m2: Subjects were treated in 21-day cycles with AB-16B5 at a dose of 12 mg/kg once weekly on Days 1, 8 and 15 combined with docetaxel at a dose of 75 mg/m2 on Day 1. Study treatment continued until there was evidence of disease progression, unacceptable toxicity, withdrawal of consent or the Investigator felt that further treatment was not in the subject's best interest, whichever occurred first.
Period: Overall Study
Arm/Group | AB-16B5 12 mg/kg & Docetaxel 75 mg/m2
Started | 35
Completed (As per protocol, study treatment continued until there was evidence of disease progression, unacceptable toxicity, withdrawal of consent or the Investigator felt that further treatment was not in the subject's best interest, whichever occurred first. Since there was no pre-defined study duration, none of the subjects is considered to have completed the study.) | 0
Not Completed | 35
Not completed — Disease Progression | 20
Not completed — Adverse Event | 5
Not completed — Physician Decision | 4
Not completed — Death | 3
Not completed — Other | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | AB-16B5 12 mg/kg & Docetaxel 75 mg/m2
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (9.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 31
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  Canada | 26
  United States | 9
Histological Classification of NSCLC [Count of Participants; unit: Participants]
  Adenocarcinoma | 28
  Squamous Cell Lung Cancer | 6
  Adenosquamous | 1
Eastern Cooperative Oncology Group (ECOG) Score [Count of Participants; unit: Participants] — The ECOG Performance Status Scale describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability.
  0. Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  Participants
    0 | 11
    1 | 22
    2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Objective response rate (ORR) was defined as the percent of subjects documented to have a confirmed complete response (CR) or partial response (PR) as per RECIST 1.1 where Complete Response (CR): disappearance of all target lesions; Partial Response (PR): at least a 30% decrease in the sum of diameters of target lesions.
Time Frame: Every 6 weeks until the date of objectively documented progression for up to 2 years.
Population: In accordance with the Statistical Analysis Plan, the analysis population for the endpoint Objective Response Rate was the Clinical Activity Evaluable (CAE) population which included all subjects who received at least one dose of each study treatment drug (AB-16B5 and Docetaxel) and who had at least one on-study disease assessment (post-dose) or developed early progression and discontinued study treatment prior to the first planned on-study disease assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | AB-16B5 12 mg/kg & Docetaxel 75 mg/m2
Number analyzed (Participants) | 35
Participants | 6

2. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: Clinical benefit rate (CBR) was defined as the percentage of subjects with complete response (CR), partial response (PR) or stable disease (SD) as per RECIST 1.1 where Complete Response (CR): disappearance of all target lesions; Partial Response (PR): at least a 30% decrease in the sum of diameters of target lesions; Stable Disease (SD): neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: Every 6 weeks until the date of objectively documented progression for up to 2 years.
Population: In accordance with the Statistical Analysis Plan, the analysis population for the endpoint Clinical Benefit Rate was the Clinical Activity Evaluable (CAE) population which included all subjects who received at least one dose of each study treatment drug (AB-16B5 and Docetaxel) and who had at least one on-study disease assessment (post-dose) or developed early progression and discontinued study treatment prior to the first planned on-study disease assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | AB-16B5 12 mg/kg & Docetaxel 75 mg/m2
Number analyzed (Participants) | 35
Participants | 16

3. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response (DOR) was defined as the time from date of the first documentation of objective tumor response (CR or PR) to the first documentation of objective progression of disease (PD) as per RECIST 1.1 or to death due to any cause in the absence of documented PD. DOR was calculated only for the subjects achieving a confirmed CR or PR. As per RECIST 1.1, Complete Response (CR): disappearance of all target lesions; Partial Response (PR): at least a 30% decrease in the sum of diameters of target lesions; Progressive Disease (PD): at least a 20% increase in the sum of diameters of target lesions, or the appearance of one or more new lesions.
Time Frame: Every 6 weeks until the date of objectively documented progression for up to 2 years.
Population: In accordance with the Statistical Analysis Plan, the analysis population for the endpoint Duration of Response was the subjects achieving a confirmed CR or PR and who received at least one dose of each study treatment drug (AB-16B5 and Docetaxel).
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | AB-16B5 12 mg/kg & Docetaxel 75 mg/m2
Number analyzed (Participants) | 6
Days | 283.50 [81.00 to 548.00]

4. Secondary Outcome: Duration of Clinical Benefit
Description: Duration of clinical benefit (CB) was defined as the time from date of the first documentation of clinical benefit (either CR, PR or SD) to the first documentation of objective progression of disease (PD) as per RECIST 1.1 or to death due to any cause in the absence of documented PD. Duration of clinical benefit was calculated only for the subjects achieving a clinical benefit. As per RECIST 1.1, Complete Response (CR): disappearance of all target lesions; Partial Response (PR): at least a 30% decrease in the sum of diameters of target lesions; Stable Disease (SD): neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD; Progressive Disease (PD): at least a 20% increase in the sum of diameters of target lesions, or the appearance of one or more new lesions.
Time Frame: Every 6 weeks until the date of objectively documented progression for up to 2 years.
Population: In accordance with the Statistical Analysis Plan, the analysis population for the endpoint Duration of Clinical Benefit was the subjects achieving a clinical benefit (either CR, PR or SD) and who received at least one dose of each study treatment drug (AB-16B5 and Docetaxel).
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | AB-16B5 12 mg/kg & Docetaxel 75 mg/m2
Number analyzed (Participants) | 16
Days | 230.00 [108.00 to 447.00]

5. Secondary Outcome: Duration of Stable Disease
Description: Duration of stable disease (SD) was defined as the time from the date of the first study treatment to the first documentation of objective progression of disease (PD) as per RECIST 1.1 or to death due to any cause in the absence of documented PD. Duration of stable disease was calculated only for the subjects achieving a stable disease as their best overall response. The best overall response was defined as the best response recorded from the start of the study treatment until the end of study. As per RECIST 1.1, Stable Disease (SD): neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD; Progressive Disease (PD): at least a 20% increase in the sum of diameters of target lesions, or the appearance of one or more new lesions.
Time Frame: Every 6 weeks until the date of objectively documented progression for up to 2 years.
Population: In accordance with the Statistical Analysis Plan, the analysis population for the endpoint Duration of Stable Disease was the subjects achieving a stable disease as their best overall response and who received at least one dose of each study treatment drug (AB-16B5 and Docetaxel).
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | AB-16B5 12 mg/kg & Docetaxel 75 mg/m2
Number analyzed (Participants) | 10
Days | 255.00 [128.00 to 543.00]

6. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression-free survival (PFS) was defined as the time from the date of first study treatment to the first documentation of objective progression of disease (PD) as per RECIST 1.1 or to death due to any cause in the absence of documented PD. For subjects who remained alive without progression at the end of the study, the event date was censored at the date of last disease assessment.
  As per RECIST 1.1, Progressive Disease (PD): at least a 20% increase in the sum of diameters of target lesions, or the appearance of one or more new lesions.
Time Frame: Every 6 weeks until the date of objectively documented progression for up to 2 years.
Population: In accordance with the Statistical Analysis Plan, the analysis population for the endpoint of Progression-free Survival was the modified Intent-to-Treat (mITT) population which included subjects who received at least one dose of each study treatment (AB-16B5 and Docetaxel).
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | AB-16B5 12 mg/kg & Docetaxel 75 mg/m2
Number analyzed (Participants) | 35
Days | 118.00 [47.00 to 231.00]

7. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) was defined as the time from date of first study treatment to death due to any cause. For surviving subjects at the end of the study, the OS endpoint was censored at the date of last contact (or last date known to be alive).
Time Frame: From the start of study treatment up to the date of death or date of last contact for up to 3 years.
Population: In accordance with the Statistical Analysis Plan, the analysis population for the endpoint Overall Survival was the modified Intent-to-Treat (mITT) population which included subjects who received at least one dose of each study treatment (AB-16B5 and Docetaxel).
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | AB-16B5 12 mg/kg & Docetaxel 75 mg/m2
Number analyzed (Participants) | 35
Days | 234.00 [148.00 to 437.00]

ADVERSE EVENTS:
Time Frame: For up to 3 years.
Description: All-cause mortality includes deaths that occurred during study treatment period and survival follow-up.
  Treatment-emergent adverse events (TEAE) are defined as any event that begins or worsens after the start of protocol treatment.
Arm/Group | AB-16B5 12 mg/kg & Docetaxel 75 mg/m2
All-Cause Mortality (participants affected / at risk) | 23/35
Serious Adverse Events (participants affected / at risk) | 23/35
Other Adverse Events (participants affected / at risk) | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AB-16B5 12 mg/kg & Docetaxel 75 mg/m2 (N=35)
Pneumonia (Infections and infestations) | 7
Diverticulitis (Infections and infestations) | 2
COVID-19 (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 1
Diverticulitis intestinal perforated (Infections and infestations) | 1
Groin infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Vascular disorders) | 3
Capillary leak syndrome (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1
Disease progression (General disorders) | 2
Non-cardiac chest pain (General disorders) | 1
Pyrexia (General disorders) | 1
Vascular stent thrombosis (General disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 2
Angina pectoris (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 1
Retinopathy (Eye disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Ischaemic stroke (Nervous system disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AB-16B5 12 mg/kg & Docetaxel 75 mg/m2 (N=35)
Anaemia (Blood and lymphatic system disorders) | 16
Neutropenia (Blood and lymphatic system disorders) | 13
Neutrophilia (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Atrial fibrillation (Cardiac disorders) | 2
Tachycardia (Cardiac disorders) | 5
Vertigo (Ear and labyrinth disorders) | 3
Hypothyroidism (Endocrine disorders) | 2
Conjunctival haemorrhage (Eye disorders) | 2
Lacrimation increased (Eye disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 7
Constipation (Gastrointestinal disorders) | 8
Diarrhoea (Gastrointestinal disorders) | 16
Dyspepsia (Gastrointestinal disorders) | 3
Mouth ulceration (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 17
Rectal haemorrhage (Gastrointestinal disorders) | 2
Stomatitis (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 10
Chest pain (General disorders) | 3
Chills (General disorders) | 4
Fatigue (General disorders) | 29
Infusion site extravasation (General disorders) | 2
Injection site reaction (General disorders) | 8
Oedema (General disorders) | 3
Oedema peripheral (General disorders) | 11
Pain (General disorders) | 3
Pyrexia (General disorders) | 12
COVID-19 (Infections and infestations) | 3
Oral candidiasis (Infections and infestations) | 6
Pneumonia (Infections and infestations) | 6
Skin infection (Infections and infestations) | 4
Urinary tract infection (Infections and infestations) | 4
Fall (Injury, poisoning and procedural complications) | 3
Infusion related reaction (Injury, poisoning and procedural complications) | 16
Alanine aminotransferase increased (Investigations) | 2
Blood alkaline phosphatase increased (Investigations) | 2
Weight decreased (Investigations) | 8
Weight increased (Investigations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 12
Dehydration (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 6
Hypokalaemia (Metabolism and nutrition disorders) | 9
Hypomagnesaemia (Metabolism and nutrition disorders) | 11
Hyponatraemia (Metabolism and nutrition disorders) | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 8
Back pain (Musculoskeletal and connective tissue disorders) | 7
Bone pain (Musculoskeletal and connective tissue disorders) | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 9
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Dizziness (Nervous system disorders) | 6
Dysgeusia (Nervous system disorders) | 6
Headache (Nervous system disorders) | 9
Neuropathy peripheral (Nervous system disorders) | 6
Paraesthesia (Nervous system disorders) | 6
Somnolence (Nervous system disorders) | 4
Anxiety (Psychiatric disorders) | 3
Confusional state (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 9
Haematuria (Renal and urinary disorders) | 2
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 25
Dry skin (Skin and subcutaneous tissue disorders) | 4
Ecchymosis (Skin and subcutaneous tissue disorders) | 6
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
Nail discolouration (Skin and subcutaneous tissue disorders) | 3
Nail disorder (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 3
Flushing (Vascular disorders) | 2
Haematoma (Vascular disorders) | 3
Hypotension (Vascular disorders) | 8
Thrombophlebitis (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-30): https://cdn.clinicaltrials.gov/large-docs/20/NCT04364620/Prot_SAP_000.pdf